CLINICAL TRIAL: NCT02794480
Title: 204980: An Open-label Study to Evaluate the Correct Use of Placebo ELLIPTA™ Dry Powder Inhaler (DPI) Compared to Placebo Metered Dose Inhalers (MDI) in Subjects With Moderate Persistent Asthma
Brief Title: Phase IV Study in Asthma Subjects for Dry Powder Inhaler (DPI) Versus (vs) Metered Dose Inhaler (MDI) Correct Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 204980
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Results first posted 2018-03-16 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Asthma
Keywords: ELLIPTA; metered dose inhaler; Dry powder inhaler
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo ELLIPTA DPI (QD) in P1 and Placebo AZ MDI (BD) in P2 (Experimental): Eligible subject will receive ELLIPTA DPI taken as one inhalation once daily (QD) for 28 days and Placebo AZ MDI taken as two inhalations twice daily (BD) for next 28 days. Subject will continue to take asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period
  Interventions: Device: ELLIPTA DPI; Device: AZ MDI
- Placebo AZ MDI (BD) in P1 and Placebo ELLIPTA DPI (QD) in P2 (Experimental): Eligible subject will receive AZ MDI taken as two inhalations twice daily for 28 days and Placebo ELLIPTA DPI taken as one inhalation once daily for next 28 days. Subject will continue to take asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period
  Interventions: Device: ELLIPTA DPI; Device: AZ MDI
- Placebo ELLIPTA DPI (QD) in P1 and Placebo GSK MDI (BD) in P2 (Experimental): Eligible subject will receive ELLIPTA DPI taken as one inhalation once daily for 28 days and Placebo GSK MDI taken as two inhalations twice daily for next 28 days. Subject will continue to take asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period.
  Interventions: Device: ELLIPTA DPI; Device: GSK MDI
- Placebo GSK MDI (BD) in P1 and Placebo ELLIPTA DPI (QD) in P2 (Experimental): Eligible subject will receive GSK MDI taken as two inhalations twice daily for 28 days and Placebo ELLIPTA DPI taken as one inhalation once daily for next 28 days. Subject will continue to take asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period
  Interventions: Device: ELLIPTA DPI; Device: GSK MDI

INTERVENTIONS:
Device: ELLIPTA DPI — It is the inhaler with two blister strips containing white coloured powder, one placebo strip containing lactose monohydrate and a second placebo strip containing lactose monohydrate blended with magnesium stearate. It is given as oral inhalation (Inhalation powder)
Device: GSK MDI — It is the placebo inhaler with clear liquid containing propellant (1,1,1, 2- Tetrafluoroethane). It is given as oral inhalation (Inhalation Aerosol).
  Arms: Placebo ELLIPTA DPI (QD) in P1 and Placebo GSK MDI (BD) in P2; Placebo GSK MDI (BD) in P1 and Placebo ELLIPTA DPI (QD) in P2
Device: AZ MDI — It is the placebo inhaler with clear liquid. It is given as oral inhalation (Inhalation Aerosol).
  Arms: Placebo AZ MDI (BD) in P1 and Placebo ELLIPTA DPI (QD) in P2; Placebo ELLIPTA DPI (QD) in P1 and Placebo AZ MDI (BD) in P2

SUMMARY:
The study is conducted to evaluate the potentially improved patient handling of the ELLIPTA Dry Powder Inhaler (DPI). Therefore, the study aims to evaluate errors encountered by subject with asthma during handling ELLIPTA DPI relative to two metered dose inhalers (MDI), a GSK MDI and the AstraZeneca (AZ) MDI. It is a randomised, multi-centre, open-label, cross-over study comparing placebo ELLIPTA DPI with placebo MDI (GSK and AZ) to assess correct inhaler use. No active drug will be used in this study in order to prevent any drug-related effects. Approximately, 152 subjects will be randomized to receive ELLIPTA DPI inhaler and 152 will be randomized to receive one of the MDI inhalers, for use during the first period (P) (approximately 28 days). At Visit 2 (Day 28) all subjects previous receiving the ELLIPTA DPI will be randomized to receive one of the MDI inhalers and all subjects who received a MDI in the previous period will receive the ELLIPTA DPI for use during second period (approximately 28 days). Subjects will continue taking their asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period.

ELLIPTA is a registered trademark of the GSK group of companies.

ELIGIBILITY:
Inclusion Criteria:

* - Subjects aged 18 years or older, at the time of signing the informed consent
* Documented history of moderate persistent asthma
* Asthma Control Test (ACT) score >=20
* Male or Females (who are not pregnant or planning pregnancy during the study or not lactating)
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions
* Subject understands and is willing, able, and likely to comply with study procedures and restrictions
* Subject must be able to read, comprehend, and record information in English
* Should not have received maintenance therapy via MDI or ELLIPTA in the past six months (DISKUS (trade name owned by GSK group of companies under license), TWISTHALER (trade name owned by Merck Sharp & Dohme Corporation, a subsidiary of Merck & Co, under license, etc are acceptable). Subject must be on maintenance therapy for 3 months, have not changed dose in the month prior to inclusion and be able to continue using their maintenance therapy throughout the study
* Requires Short-acting-beta-agonist (SABA) for symptom control =<2 days/week. Use of SABA prior to exercise for the prevention of exercise induced bronchoconstriction is exclusionary.

Exclusion Criteria:

* Subjects with a known or suspected alcohol or drug abuse at Visit 1 which in the opinion of the investigator could interfere with the subject's proper completion of the protocol requirement
* Current smokers or subjects with a smoking history of 10 pack-years or more (example, 20 cigarettes/day for 10 years) are not eligible. A subject may not have used tobacco products within the past year (i.e., cigarettes, cigars, or pipe tobacco)
* Concurrent diagnosis of chronic obstructive pulmonary disease (COPD) or other respiratory disorders including active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases
* History of life threatening asthma or has experienced more than 1 exacerbation which required oral/systemic corticosteroids in the 12 months prior to Visit 1
* History of hypersensitivity to any components of the study inhaler (e.g., lactose, magnesium stearate). In addition, subjects with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates participation
* Historical or current evidence of clinically significant or rapidly progressing or unstable cardiovascular, neurological, cardiovascular, neurological, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the affect the analysis if the disease/condition exacerbated during the study
* Subjects who have received an investigational drug and/or medical device within 30 days of entry into this study (Screening/Visit 1), or within five drug half-lives of the investigational drug, whichever is longer
* A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- United States (20):
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, Warrensburg, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=204980

REFERENCES:
- [Background] Kerwin EM, Preece A, Brintziki D, Collison KA, Sharma R. ELLIPTA Dry Powder Versus Metered-Dose Inhalers in an Optimized Clinical Trial Setting. J Allergy Clin Immunol Pract. 2019 Jul-Aug;7(6):1843-1849. doi: 10.1016/j.jaip.2019.02.023. Epub 2019 Mar 2. PMID 30836228

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized, multi-center, open-label, cross-over study comparing Placebo ELLIPTA Dry Power Inhaler (DPI) with either Placebo GlaxoSmithKline (GSK) Metered Dose Inhaler (MDI) or Placebo Astra Zeneca (AZ) MDI to assess correct inhaler use. A total of 20 sites in the United States (US) participated in the study.
Pre-assignment Details: A total of 329 participants (par) were screened out of which 324 were randomized to sub-study 1 and sub-study 2 in a ratio of 1:1. Each par received at least one-dose of placebo from at least one study inhaler. These par comprised the intent to treat (ITT) population. Par were randomized on the same day as screening.
Groups:
- Sub-Study 1 (Seq 3: Ellipta/GSK MDI); Sub-Study 1 (Seq 4: GSK MDI/Ellipta): Par were randomized to treatment sequence 3 or 4. In treatment sequence 3, the par were dispensed Placebo ELLIPTA DPI at Visit 1 for treatment period 1 and Placebo GSK MDI at Visit 2 for treatment period 2. In treatment sequence 4, the par were dispensed Placebo GSK MDI at Visit 1 for treatment period 1 and Placebo ELLIPTA DPI at Visit 2 for treatment period 2. ELLIPTA was a two strip inhaler with one placebo strip containing lactose monohydrate and a second placebo strip containing lactose monohydrate blended with magnesium stearate. GSK MDI contained propellant (1,1,1,2-Tetrafluoroethane). ELLIPTA DPI was taken as one inhalation, once daily and GSK MDI was taken as two inhalations, twice daily. Par continued taking their asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period.
- Sub-Study 2 (Seq 1: Ellipta/AZ MDI); Sub-Study 2 (Seq 2: AZ MDI/Ellipta): Par were randomized to treatment sequence 1 or 2. In treatment sequence 1, the par were dispensed Placebo ELLIPTA DPI at Visit 1 for treatment period 1 and Placebo AZ MDI at Visit 2 for treatment period 2. In treatment sequence 2, the par were dispensed Placebo AZ MDI at Visit 1 for treatment period 1 and Placebo ELLIPTA DPI at Visit 2 for treatment period 2. ELLIPTA was a two strip inhaler with one placebo strip containing lactose monohydrate and a second placebo strip containing lactose monohydrate blended with magnesium stearate. AZ MDI was a placebo inhaler containing liquid aerosol. ELLIPTA DPI was taken as one inhalation, once daily and AZ MDI was taken as two inhalations, twice daily. Par continued taking their asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period.
Period: Period 1: Treatment Period 1 (28 Days)
Arm/Group | Sub-Study 1 (Seq 3: Ellipta/GSK MDI) | Sub-Study 1 (Seq 4: GSK MDI/Ellipta) | Sub-Study 2 (Seq 1: Ellipta/AZ MDI) | Sub-Study 2 (Seq 2: AZ MDI/Ellipta)
Started | 80 | 82 | 81 | 81
Completed | 80 | 80 | 79 | 78
Not Completed | 0 | 2 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1
Period: Period 2: Treatment Period 2 (28 Days)
Arm/Group | Sub-Study 1 (Seq 3: Ellipta/GSK MDI) | Sub-Study 1 (Seq 4: GSK MDI/Ellipta) | Sub-Study 2 (Seq 1: Ellipta/AZ MDI) | Sub-Study 2 (Seq 2: AZ MDI/Ellipta)
Started | 80 | 80 | 79 | 78
Completed | 79 | 80 | 79 | 77
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sub-Study 1 (Seq 3: Ellipta/GSK MDI; Seq 4: GSK MDI/Ellipta): Par were randomized to treatment sequence 3 or 4. In treatment sequence 3, the par were dispensed Placebo ELLIPTA DPI at Visit 1 for treatment period 1 and Placebo GSK MDI at Visit 2 for treatment period 2. In treatment sequence 4, the par were dispensed Placebo GSK MDI at Visit 1 for treatment period 1 and Placebo ELLIPTA DPI at Visit 2 for treatment period 2. ELLIPTA was a two strip inhaler with one placebo strip containing lactose monohydrate and a second placebo strip containing lactose monohydrate blended with magnesium stearate. GSK MDI contained propellant (1,1,1,2-Tetrafluoroethane). ELLIPTA DPI was taken as one inhalation, once daily and GSK MDI was taken as two inhalations, twice daily. Par continued taking their asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period.
- Sub-Study 2 (Seq 1: Ellipta/AZ MDI; Seq 2: AZ MDI/Ellipta): Par were randomized to treatment sequence 1 or 2. In treatment sequence 1, the par were dispensed Placebo ELLIPTA DPI at Visit 1 for treatment period 1 and Placebo AZ MDI at Visit 2 for treatment period 2. In treatment sequence 2, the par were dispensed Placebo AZ MDI at Visit 1 for treatment period 1 and Placebo ELLIPTA DPI at Visit 2 for treatment period 2. ELLIPTA was a two strip inhaler with one placebo strip containing lactose monohydrate and a second placebo strip containing lactose monohydrate blended with magnesium stearate. AZ MDI was a placebo inhaler containing liquid aerosol. ELLIPTA DPI was taken as one inhalation, once daily and AZ MDI was taken as two inhalations, twice daily. Par continued taking their asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period.
- Total: Total of all reporting groups
Arm/Group | Sub-Study 1 (Seq 3: Ellipta/GSK MDI; Seq 4: GSK MDI/Ellipta) | Sub-Study 2 (Seq 1: Ellipta/AZ MDI; Seq 2: AZ MDI/Ellipta) | Total
Number analyzed (Participants) | 157 | 153 | 310
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.4 (15.87) | 50.9 (15.08) | 51.1 (15.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 108 | 216
  Male | 49 | 45 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  race customized: AMERICAN INDIAN OR ALASKA NATIVE | 1 | 2 | 3
  race customized: ASIAN - CENTRAL/SOUTH ASIAN HERITAGE | 1 | 0 | 1
  race customized: ASIAN - EAST ASIAN HERITAGE | 0 | 1 | 1
  race customized: ASIAN - JAPANESE HERITAGE | 1 | 0 | 1
  race customized: ASIAN - SOUTH EAST ASIAN HERITAGE | 2 | 1 | 3
  race customized: BLACK OR AFRICAN AMERICAN | 36 | 33 | 69
  race customized: WHITE - ARABIC/NORTH AFRICAN HERITAGE | 0 | 1 | 1
  race customized: WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | 115 | 113 | 228
  race customized: MULTIPLE | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Zero Errors in ELLIPTA DPI Versus GSK MDI and AZ MDI After 28 Days of Use in Each Treatment Phase
Description: A checklist for correct use of each inhaler was developed based on the steps identified in the package insert. Baseline assessment was conducted when the par were dispensed the inhaler and were guided by a trained healthcare provider (HCP) to demonstrate correct use of the assigned inhaler. A second assessment was conducted after each 28 day dosing period without instruction by HCP. The Correct Use Check list was completed by HCP at each visit. Percentage of par with zero errors in inhaler use at Day 28, was analyzed using a Mainland-Gart test for each ELLIPTA versus MDI comparison separately (Sub-study 1: ELLIPTA vs GSK MDI and Sub-study 2: ELLIPTA vs AZ MDI). For each ELLIPTA vs MDI analyses, only par who made no error in any of the inhalers and at least one error on the other inhaler (discordant cases) were included in the analysis. NA indicates that par did not receive the inhaler in that particular sub-study.
Time Frame: Up to Day 56
Population: Modified ITT Population (MITT) comprises of all par in the ITT Population who provided Day 28 inhaler use data for both of their randomized inhalers.
Measure: Number; unit: Percentage of Participants
Groups:
- Sub-Study 1: Par were randomized to treatment sequence 3 or 4. In treatment sequence 3, the par were dispensed Placebo ELLIPTA DPI at Visit 1 for treatment period 1 and Placebo GSK MDI at Visit 2 for treatment period 2. In treatment sequence 4, the par were dispensed Placebo GSK MDI at Visit 1 for treatment period 1 and Placebo ELLIPTA DPI at Visit 2 for treatment period 2. ELLIPTA was a two strip inhaler with one placebo strip containing lactose monohydrate and a second placebo strip containing lactose monohydrate blended with magnesium stearate. GSK MDI contained propellant (1,1,1,2-Tetrafluoroethane). ELLIPTA DPI was taken as one inhalation, once daily and GSK MDI was taken as two inhalations, twice daily. Par continued taking their asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period.
- Sub-Study 2: Par were randomized to treatment sequence 1 or 2. In treatment sequence 1, the par were dispensed Placebo ELLIPTA DPI at Visit 1 for treatment period 1 and Placebo AZ MDI at Visit 2 for treatment period 2. In treatment sequence 2, the par were dispensed Placebo AZ MDI at Visit 1 for treatment period 1 and Placebo ELLIPTA DPI at Visit 2 for treatment period 2. ELLIPTA was a two strip inhaler with one placebo strip containing lactose monohydrate and a second placebo strip containing lactose monohydrate blended with magnesium stearate. AZ MDI was a placebo inhaler containing liquid aerosol. ELLIPTA DPI was taken as one inhalation, once daily and AZ MDI was taken as two inhalations, twice daily. Par continued taking their asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period.
Arm/Group | Sub-Study 1 | Sub-Study 2
Number analyzed (Participants) | 24 | 15
Percentage of Participants
  ELLIPTA | 87 | 87
  GSK MDI | 13 | NA — NA indicates that the par did not receive the inhaler in that particular sub-study.
  AZ MDI | NA — NA indicates that the par did not receive the inhaler in that particular sub-study. | 13
Statistical Analysis 1: Comparison: Sub-Study 1; Test type: Superiority; p < 0.001, Mainland-Gart test — ELLIPTA versus GSK MDI; Mainland-Gart test is favorable over the McNemar test for matched pairs as the latter is only valid in case of no period effects
Statistical Analysis 2: Comparison: Sub-Study 2; Test type: Superiority; p = 0.007, Mainland-Gart test — ELLIPTA versus AZ MDI; [other analysis details as in outcome 1, analysis 1]

2. Secondary Outcome: Frequency of Errors by Type for ELLIPTA After 28 Days of Use in Each Treatment Phase
Description: The occurrence of each type of error while using ELLIPTA inhaler was evaluated based on the information collected in the Correct Use Checklists. The number of errors for each type of inhaler was assessed at Visit 2 and Visit 3. The par were counted more than once depending on the reasons for incorrect use. Only par who made at least one error was included in the summary (represented by the number of Participants).
Time Frame: Up to Day 56
Population: MITT Population
Measure: Number; unit: Participants
Arm/Group | Sub-Study 1 | Sub-Study 2
Number analyzed (Participants) | 7 | 3
Participants
  Par did shake the inhaler (ir) | 3 | 0
  Par didn't exhale when ir was held away from mouth | 2 | 2
  Par breathed into the mouthpiece (mp) | 2 | 0
  Mp was not placed with lips closed around it | 1 | 0
  Par did not take one long steady deep breath | 1 | 1
  Par didn't remove ir from mouth and hold breath | 1 | 1
  Par did not breathe out slowly and gently | 1 | 2

3. Secondary Outcome: Frequency of Errors by Type for MDI After 28 Days of Use in Each Treatment Phase
Description: The occurrence of each type of error while using GSK MDI in Sub-Study 1 and AZ MDI in Sub-Study 2 was evaluated based on the information collected in the Correct Use Checklists. The number of errors for each type of inhaler was assessed at Visit 2 and Visit 3. The par were counted more than once depending on the reasons for incorrect use. The number of errors is reported as NA for the type of error which was not applicable to the particular inhaler type. Only par who made at least one error are included in the summary (represented by the number of Participants).
Time Frame: Up to Day 56
Population: MITT Population
Measure: Number; unit: Participants
Arm/Group | Sub-Study 1 | Sub-Study 2
Number analyzed (Participants) | 25 | 14
Participants
  Par did not shake the inhaler | 5 | 5
  Par did not check the mp for foreign objects | 14 | 9
  Par did not hold the inhaler with the mp down | 1 | NA — The number of errors are reported as NA for the type of error which was not applicable to the particular inhaler type.
  Par did not breathe out fully | 5 | 0
  Mp was not placed with lips closed around it | 2 | 0
  Par did not press top of canister all way down | 2 | 2
  Ability to release actuation was not demonstrated | 4 | 2
  Par did not take finger off the canister | 3 | 2
  Par did not remove inhaler from mouth & closed it | 2 | NA — The number of errors are reported as NA for the type of error which was not applicable to the particular inhaler type.
  Par didn't hold breath for 10 s & exhale slowly | 3 | 2
  Par did not snap the cap back firmly into place | 2 | 0
  Inhaler was not kept upright & removed from mouth | NA — The number of errors are reported as NA for the type of error which was not applicable to the particular inhaler type. | 2
  Par did not close the inhaler completely | NA — The number of errors are reported as NA for the type of error which was not applicable to the particular inhaler type. | 1

4. Secondary Outcome: Number of Errors Per Participant for Each Inhaler After 28 Days of Use (All Evaluable Par)
Description: The number of errors per par for each inhaler (ELLIPTA and GSK MDI or AZ MDI) was evaluated based on the information collected in the Correct Use Checklists. The number of errors per par was summarised as continuous data by inhaler for each of the ELLIPTA versus MDI comparisons. NA indicates that the par did not receive the inhaler in that particular sub-study.
Time Frame: Up to Day 56
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | Sub-Study 1 | Sub-Study 2
Number analyzed (Participants) | 157 | 153
Errors
  ELLIPTA | 0.07 (0.393) | 0.04 (0.299)
  GSK MDI | 0.35 (1.139) | NA (NA) — NA indicates that the par did not receive the inhaler in that particular study.
  AZ MDI | NA (NA) — NA indicates that the par did not receive the inhaler in that particular study. | 0.21 (0.838)

5. Secondary Outcome: Number of Errors Per Participant for Each After 28 Days of Use (Par With at Least One Error)
Description: The number of errors for each inhaler (ELLIPTA and GSK MDI or AZ MDI) in par with one or more errors were evaluated based on the information collected in the Correct Use Checklists. The number of errors per par was summarised as continuous data by inhaler for each of the ELLIPTA versus MDI comparisons. NA indicates that the par. did not receive the inhaler in that particular sub-study. Only those par who made at least one error were included in the summary (represented by n=X, X in the category titles).
Time Frame: Up to Day 56
Population: MITT Population
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | Sub-Study 1 | Sub-Study 2
Number analyzed (Participants) | 157 | 153
Errors
  ELLIPTA; n=7, 3: number analyzed (Participants) | 7 | 3
  ELLIPTA; n=7, 3 | 1.57 (1.134) | 2.00 (1.000)
  GSK MDI; n=25, 0: number analyzed (Participants) | 25 | 0
  GSK MDI; n=25, 0 | 2.20 (2.062) |
  AZ MDI; n=0, 14: number analyzed (Participants) | 0 | 14
  AZ MDI; n=0, 14 |  | 2.29 (1.773)

6. Post Hoc Outcome: Percentage of Participants With Zero Errors in ELLIPTA DPI Versus GSK MDI and AZ MDI After 28 Days of Use in Each Treatment Phase
Description: A supportive post-hoc analysis on the primary endpoint was performed to address possible concerns due to the exclusion of data from a large number of participants who made no errors or at least one error on either inhaler tested in the primary analysis (only discordant cases involved in the analysis). For each ELLIPTA versus MDI comparison separately (Sub-study 1: Ellipta vs GSK MDI and Sub-study 2: Ellipta vs AZ MDI), the percentage of par having zero errors in inhaler use at Day 28 was analyzed using a Conditional Logistic Regression adjusting for treatment (inhaler) and treatment period. NA indicates that the par did not receive the inhaler in that particular sub-study.
Time Frame: Up to Day 56
Population: MITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Sub-Study 1 | Sub-Study 2
Number analyzed (Participants) | 157 | 153
Percentage of Participants
  Zero Errors after 28 Days of Use ELLIPTA | 96 | 98
  Zero Errors after 28 Days of Use GSK MDI | 84 | NA — NA indicates that the par. did not receive the inhaler in that particular sub-study.
  Zero Errors after 28 Days of Use AZ MDI | NA — NA indicates that the par. did not receive the inhaler in that particular sub-study. | 91
  At least one Error after 28 Days of Use ELLIPTA | 4 | 2
  At least one Error after 28 Days of Use GSK MDI | 16 | NA — NA indicates that the par. did not receive the inhaler in that particular sub-study.
  At least one Error after 28 Days of Use AZ MDI | NA — NA indicates that the par. did not receive the inhaler in that particular sub-study. | 9
Statistical Analysis 1: Comparison: Sub-Study 1; Test type: Superiority; p < 0.001, Conditional Logistic Regression — Exact odds ratio calculated using exact conditional logistic regression adjusted for treatment and treatment period; Odds Ratio (OR) = 5.94, 95% CI 2-sided [lower limit 2.42] (The upper limit is infinity.) — ELLIPTA versus GSK MDI
Statistical Analysis 2: Comparison: Sub-Study 2; Test type: Superiority; p = 0.011, Conditional Logistic Regression — Exact odds ratio calculated using exact conditional logistic regression adjusted for treatment and treatment period; Odds Ratio (OR) = 4.16, 95% CI 2-sided [lower limit 1.59] (The upper limit is infinity.) — ELLIPTA versus AZ MDI

ADVERSE EVENTS:
Time Frame: On-treatment adverse events (AEs) and serious adverse events (SAEs) were collected from the start of study treatment and until the follow up visit (up to 58 days).
Description: On-treatment AEs and SAEs were reported for ITT population.
Groups:
- Sub-Study 1 - Ellipta (Sequence 3,4); Sub-Study 1 - GSK MDI (Sequence 3,4): Par were randomized to treatment sequence 3 or 4. In treatment sequence 3, the par were dispensed Placebo ELLIPTA DPI at Visit 1 for treatment period 1 and Placebo GSK MDI at Visit 2 for treatment period 2. In treatment sequence 4, the par were dispensed Placebo GSK MDI at Visit 1 for treatment period 1 and Placebo ELLIPTA DPI at Visit 2 for treatment period 2. ELLIPTA was a two strip inhaler with one placebo strip containing lactose monohydrate and a second placebo strip containing lactose monohydrate blended with magnesium stearate. GSK MDI contained propellant (1,1,1,2-Tetrafluoroethane). ELLIPTA DPI was taken as one inhalation, once daily and GSK MDI was taken as two inhalations, twice daily. Par continued taking their asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period.
- Sub-Study 2 - Ellipta (Sequence 1,2); Sub-Study 2 - AZ MDI (Sequence 1,2): Par were randomized to treatment sequence 1 or 2. In treatment sequence 1, the par were dispensed Placebo ELLIPTA DPI at Visit 1 for treatment period 1 and Placebo AZ MDI at Visit 2 for treatment period 2. In treatment sequence 2, the par were dispensed Placebo AZ MDI at Visit 1 for treatment period 1 and Placebo ELLIPTA DPI at Visit 2 for treatment period 2. ELLIPTA was a two strip inhaler with one placebo strip containing lactose monohydrate and a second placebo strip containing lactose monohydrate blended with magnesium stearate. AZ MDI was a placebo inhaler containing liquid aerosol. ELLIPTA DPI was taken as one inhalation, once daily and AZ MDI was taken as two inhalations, twice daily. Par continued taking their asthma maintenance treatment and limited rescue albuterol MDI during the entire 56-day study period.
Arm/Group | Sub-Study 1 - Ellipta (Sequence 3,4) | Sub-Study 1 - GSK MDI (Sequence 3,4) | Sub-Study 2 - Ellipta (Sequence 1,2) | Sub-Study 2 - AZ MDI (Sequence 1,2)
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/162 | 0/162 | 0/162
Serious Adverse Events (participants affected / at risk) | 0/162 | 0/162 | 0/162 | 0/162
Other Adverse Events (participants affected / at risk) | 12/162 | 16/162 | 15/162 | 17/162
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sub-Study 1 - Ellipta (Sequence 3,4) (N=162) | Sub-Study 1 - GSK MDI (Sequence 3,4) (N=162) | Sub-Study 2 - Ellipta (Sequence 1,2) (N=162) | Sub-Study 2 - AZ MDI (Sequence 1,2) (N=162)
Bronchitis (Infections and infestations) | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 2
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 1 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Sinus operation (Surgical and medical procedures) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Angular cheilitis (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0
Multiple allergies (Immune system disorders) | 0 | 0 | 0 | 1
Product taste abnormal (Product Issues) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.